CLINICAL TRIAL: NCT00638651
Title: Topical Imiquimod in Conjunction With Nd:YAG Laser for Tattoo Removal
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Graceway Pharmaceuticals, LLC (Industry)
Responsible Party: Principal Investigator, Keyvan Nouri, MD, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 20071234
Record Dates: First submitted 2008-03-12; First posted 2008-03-19 (Estimated); Results first posted 2014-09-01 (Estimated); Last update posted 2018-03-22 (Actual); Status verified 2018-02

CONDITIONS: Healthy
Keywords: Tattoos; Black/blue tattoos
MeSH Terms: interventions — Imiquimod

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): The tattoo will be treated with laser and imiquimod 5% cream
  Interventions: Device: 1064 nm Nd:YAG laser; Drug: Imiquimod, 5% cream
- 2 (Placebo Comparator): The tattoo will be treated with laser and placebo topical cream
  Interventions: Device: 1064 nm Nd:YAG laser

INTERVENTIONS:
Device: 1064 nm Nd:YAG laser — The laser used will be a 1064 nm Nd:YAG, with a 10ns pulse, 3mm spot size and 4 joules of energy
Drug: Imiquimod, 5% cream — 2 weeks after the laser procedure the imiquimod will be applied 3 times a week for one month
  Other Names: Aldara
  Arms: 1

SUMMARY:
The purpose of this study is to evaluate the efficacy of tattoo removal using topical imiquimod, 5% cream in conjunction with the 1064nm Nd:YAG laser. This procedure for tattoo removal will be compared to a laser removal alone.

DETAILED DESCRIPTION:
Inclusion criteria includes: patients of both genders with Fitzpatrick skin types I-IV who are 18-65 years of age and who has 2 tattoos from 2 to 10 cm in diameter, of similar age which contains black and/or blue ink in areas that can be covered. Exclusion criteria includes: tattoos in chronically sun exposed areas, larger than 25 cm2,pregnancy,breast feeding state, immunosuppressed patients, history of autoimmune or connective tissue disorders, hypersensitivity to imiquimod, active sunburn, current tan, use of coumadin, aspirin , vitamin E or non-steroidal anti-inflammatory agents for the past 10 days.

ELIGIBILITY:
Inclusion Criteria:

* 2 tattoos no larger than 25cm2, professionally made, with approximately the same age, containing blue/black ink.

Exclusion Criteria:

* Hypersensitivity to imiquimod
* Current sun tan
* Use of vitamin E, non-steroid anti-inflammatory drugs, coumadin or aspirin for the past 10 days
* Amateur tattoos
* Pregnancy
* Breast-feeding status
* Immunosuppression
* Auto-immune diseases.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2008-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keyvan Nouri, MD, Principal Investigator — University of Miami
Locations (1):
- Mohs, Dermatologic and Laser Surgery, Miami, Florida, United States

REFERENCES:
- [Result] Elsaie ML, Nouri K, Vejjabhinanta V, Rivas MP, Villafradez-Diaz LM, Martins A, Rosso R. Topical imiquimod in conjunction with Nd:YAG laser for tattoo removal. Lasers Med Sci. 2009 Nov;24(6):871-5. doi: 10.1007/s10103-009-0709-9. Epub 2009 Jul 15. PMID 19597914
- See also: Principal investigator biography — https://link.springer.com/article/10.1007%2Fs10103-009-0709-9

RESULTS

PARTICIPANT FLOW:
Groups:
- Laser Treatment With Imiquimod Cream or Placebo: Participants with two tattoos were selected. Each tattoo were treated with either laser and imiquimod 5% cream or laser and placebo cream.
Period: Overall Study
Arm/Group | Laser Treatment With Imiquimod Cream or Placebo
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Laser Treatment With Imiquimod Cream or Placebo: One participant with two tattoos were selected. Each tattoo were treated with either laser and imiquimod 5% cream or laser and placebo cream.
Arm/Group | Laser Treatment With Imiquimod Cream or Placebo
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of Tattoo Removal Using Topical Imiquimod 5% Cream
Description: To evaluate the efficacy of tattoo removal using topical imiquimod, 5% cream (Aldara™, 3M/Graceway Pharmaceuticals, an immune response modifier) in conjunction with the 1064 nm Nd:YAG laser. This procedure for tattoo removal will be compared to laser removal alone.
Time Frame: approximately 14 weeks
Measure: Mean (Full Range); unit: percentage of tattoo pigment removed
Units Other Than Participants: Tattoo
Groups:
- Laser Treatment With Imiquimod (Group 1): The tattoo will be treated with laser and imiquimod 5% cream
  1064 nm Nd:YAG laser: The laser used will be a 1064 nm Nd:YAG, with a 10ns pulse, 3mm spot size and 4 joules of energy
  Imiquimod, 5% cream: 2 weeks after the laser procedure the imiquimod will be applied 3 times a week for one month
- Laser Treatment With Placebo Cream (Group 2): The tattoo will be treated with laser and placebo topical cream
  1064 nm Nd:YAG laser: The laser used will be a 1064 nm Nd:YAG, with a 10ns pulse, 3mm spot size and 4 joules of energy
Arm/Group | Laser Treatment With Imiquimod (Group 1) | Laser Treatment With Placebo Cream (Group 2)
Number analyzed (Participants) | 3 | 3
Number analyzed (Tattoo) | 3 | 3
percentage of tattoo pigment removed | 4.3 [0 to 5] | 2.7 [0 to 5]

ADVERSE EVENTS:
Arm/Group | Laser Treatment With Imiquimod Cream or Placebo
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No